CLINICAL TRIAL: NCT05489029
Title: Peculiarities of Pain in Patients With Gunshot Wounds Depending on the Localization of the Wound at the Stages of Treatment
Acronym: PPPGWDL
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Chief researcher, Bogomolets National Medical University
Other Study IDs: №158/23.05.2022
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
Keywords: pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Interventions: Other: visual analog scale
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022
  Interventions: Other: visual analog scale

INTERVENTIONS:
Other: visual analog scale — Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Other Names: neuropathic pain Didier Bouhassiraa DN4; Chaban Quality of Life Scale; The Hospital Anxiety and Depression Scale (HADS); Mississippi scale of post-traumatic stress disorders (military version) (MS PTSD (m))

SUMMARY:
Chronic pain, in turn, is associated with a whole cohort of mutually aggravating factors - this can lead to the development of extremely serious long-term consequences. The features of pain in this category of patients have not been sufficiently studied. Taking into account continuity and consistency, clear and high-quality pain treatment is necessary at all stages of treatment.

DETAILED DESCRIPTION:
The peculiarities of pain in patients with gunshot wounds, depending on the localization of the wound at the stages of treatment, need to be studied, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions through the prism of psychological disorders have their own characteristics.

ELIGIBILITY:
Inclusion Criteria:

* the presence of gunshot wounds

Exclusion Criteria:

* no gunshot wounds

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: all patients were injured during hostilities
Sampling Method: Probability Sample
Enrollment: 1555 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  from 0 to 10 points
pain diagnostic questionnaire | 12 months
  4 or more points (a neuropathic pain component is present)
The Hospital Anxiety and Depression Scale | 12 months
  0-7 is the norm 8-13 - mild depressive disorders 14-18 - depressive disorders of medium severity 19-22 - severe depressive disorders 23 and more - depressive disorders of a very severe degree of severity
Chaban Quality of Life Scale | 12 months
  up to 56 inclusive - a very low level 57-66 - low 67-75 - average 76-82 - tall 83-100 is very high
Mississippi PTSD scale (military version) | 12 months
  the mean values of the total score are 76±18 for well-adjusted servicemen, 86±26 for servicemen with mental disorders, and 130±18 for those with PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share

REFERENCES:
- [Derived] Kuchyn I, Horoshko V. Chronic pain in patients with gunshot wounds. BMC Anesthesiol. 2023 Feb 7;23(1):47. doi: 10.1186/s12871-023-02005-3. PMID 36750768